CLINICAL TRIAL: NCT03703401
Title: The Role of Hydrosalpinx in Recurrent Miscarriage
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Tommy's (Other)
Responsible Party: Principal Investigator, Dr Jayasish Ghosh, Principal Investigator, University of Birmingham
Other Study IDs: IRAS ID 232650
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Abortion, Spontaneous; Miscarriage, Recurrent; Hydrosalpinx
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with recurrent miscarriage and no hydrosalpinx
  Interventions: Diagnostic Test: Hysterosalpingo-contrast-sonogram
- Women with recurrent miscarriage and concurrent hydrosalpinx
  Interventions: Diagnostic Test: Hysterosalpingo-contrast-sonogram
- Women with recurrent miscarriage and treated hydrosalpinx
  Interventions: Diagnostic Test: Hysterosalpingo-contrast-sonogram

INTERVENTIONS:
Diagnostic Test: Hysterosalpingo-contrast-sonogram — A contrast ultrasound scan to examine fallopian tube pathology and blockage

SUMMARY:
Miscarriage affects one in five pregnancies and little progress has been made in understanding and treating this distressing condition. C. trachomatis is the most common sexually transmitted infection in the UK. C. trachomatis infection can have serious health consequences, including fallopian tube damage. Untreated C. trachomatis infection and tubal damage have been associated with miscarriage and adverse pregnancy outcomes such as preterm birth, low birth weight and stillbirth. A cohort study is needed to establish the prevalence of tubal disease in women with recurrent miscarriages. HyCoSy will be performed to identify tubal disease and establish the magnitude of the problem in the recurrent miscarriage population. The prognosis of tubal disease on miscarriage and other obstetric outcomes, and the role of medical interventions such as tubal surgery (to treat hydrosalpinx) on reducing miscarriage and adverse obstetric outcomes will also be studied.

Objectives

1. Establish the prevalence of hydrosalpinx in the recurrent miscarriage population.
2. Establish the prognosis of women diagnosed with recurrent miscarriage with concurrent hydrosalpinx.
3. Explore the role of tubal surgery for improving reproductive outcomes in women with recurrent miscarriage population and hydrosalpinx.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Women diagnosed with recurrent miscarriage i.e. 2 or more miscarriages
* Ability to give informed consent

Exclusion Criteria:

* Allergy to contrast media used for Hysterosalpingo-contrast-sonogram
* Allergy to sonographic gel used for ultrasound scanning
* Anatomical anomaly meaning transvaginal ultrasound scan not possible
* Stenosed/occluded cervix meaning contrast media unable to be introduced via cervix
* Inability to give informed consent
* Pregnant at the time of recruitment
* Declined recruitment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Must be genetically female as must have suffered from previous pregnancy losses
Study Population: Women who have suffered from 2 or more pregnancy losses
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Hydrosalpinx | 12 months
  The presence or absence of tubal blockage and hydrosalpinx

SECONDARY OUTCOMES:
Miscarriage | 12 months
  The loss of a pregnancy below 24 completed week of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Womens Hospital, Birmingham, West Midands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03703401/Prot_000.pdf